CLINICAL TRIAL: NCT04025385
Title: High-Intensity-Interval-Training in Geriatric Rehabilitation - A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Michael Kruesi, Resident Physician, Doctoral Candidate, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KLV-BA-2019-1
Record Dates: First submitted 2019-06-16; First posted 2019-07-18 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Rehabilitation; Post-Operative Condition; Deconditioning After Acute Hospital; Oncology
MeSH Terms: conditions — Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients will participate in regular training units
- HIIT Group (Active Comparator): Patients will participate in high intensity interval training
  Interventions: Other: High Intensity Interval Training

INTERVENTIONS:
Other: High Intensity Interval Training — Training for 25 min with four 1 minute intervals when participants exercise up to 80% of their individual limits.
  Arms: HIIT Group

SUMMARY:
Study with Patients (40-60 participants) above the age of 65. There will be a comparison of regular training on ergometer (10 trainings within 2 weeks, 40 min each) to high intensity interval training on ergometer (6 trainings within 2 weeks, 25 min each). At the beginning and at the end will be a spiroergometer to measure the individual limits and vO2max, which will be compared amongst the two groups. To receive a subjective feedback, there will be a series of questionnaires at the beginning, after one week and at the end. The goal of this study is to get more information about whether a HII-Training is feasible with elderly patients and whether they can profit form it.

ELIGIBILITY:
Inclusion Criteria:

* cardiopulmonal resilient
* able to sit on a ergometer
* knowledge of German written and spoken

Exclusion Criteria:

* Severe cardiopulmonary restriction (LVEF <30%, conduction abnormalities from AV block IIb or higher)
* Absolute cardiopulmonary contraindications (acute coronary syndrome, unstable AP -> not capable of rehabilitation), uncompensated heart failure (dyspnea at rest, orthopnea, severe edema)
* No ischemic events (cardiac, cerebral, peripheral) within the last 3 months
* Severe pneumatological underlying disease: COPD GOLD 3 and higher or status after exacerbation within the last 2 weeks, Asthma grade 4
* Dyalisis reliant
* Severe psychiatric disorder (severe psychosis, severe depression)
* Distinct dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Will there be a change in outcome of individuals vO2max? | 2 Weeks
  Measurement of vO2max with spiroergometer at the beginning and end
Is a High intensity interval training feasible with elderly patients in rehabilitation? | 1 Day
  Questionnaire (Clinic-intern questionnaire) amongst the involved personal

SECONDARY OUTCOMES:
Will there be a change in subjective quality of life? | 2.5 Weeks
  Questionnaires (PROMIS-10, EQ-5D) amongst the participants

CONTACTS AND LOCATIONS:
Locations (1):
- Rehazentrum Walenstadtberg, Walenstadtberg, Switzerland